CLINICAL TRIAL: NCT04370626
Title: The Canadian Prospective Pragmatic Perilunate Outcomes Trial (The C3PO Trial)
Brief Title: The Canadian Prospective Pragmatic Perilunate Outcomes Trial
Acronym: C3PO
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: REB19-1565
Record Dates: First submitted 2019-10-15; First posted 2020-05-01 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-05

CONDITIONS: Wrist Injuries; Carpal Bone Fracture; Dislocation of Wrist; Trauma
MeSH Terms: conditions — Wrist Injuries; Wrist Fractures; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Registry Group: Patients who sustain and present with a PLI injury will have two options for participating in the study. This first arm will evaluate clinical presentations, patient demographic, treatment methods and baseline patient-rated and radiographic outcomes. However, no research-related follow up visits will be conducted. Ongoing data from these participants will be collected from chart reviews of clinical follow-ups alone.
- Prospective Group: Participants who choose to enroll in the prospective arm will experience the same baseline data collection as those in the registry, with the addition of research-related follow up appointments that will allow research staff to measure and assess patient-rated and clinical outcomes, such as questionnaires and range of motion data.
- Retrospective Group: In this group, a chart review will be conducted to identify previously treated patients with perilunate injuries. Once identified, the patient will be contacted and ask if they are willing to come in for a long-term follow up visit where clinical, patient-rated, and radiographic data will be collected. If patients are unwilling to attend a long-term visit, our analysis will still include data collected from their chart reviews and electronic questionnaires.

SUMMARY:
This is a unique three-fold prospective and retrospective study. With this approach, all previous and current PLIs presented at participating study sites will have the potential to be included in the study. Our goal is to collect all relevant injury and surgical parameters of the Perilunate spectrum. The investigators plan to identify each hospital within Canada that normally treats PLIs and to record injury and demographic information on each PLI that occurs in this country over a two to three-year period. Our protocol includes scheduled two, five, and 10-year follow-up intervals.

DETAILED DESCRIPTION:
Perilunate injuries commonly occur from high-energy sporting or automobile accidents and require urgent surgical intervention. Although these wrist injuries are commonly encountered in the population, their complexity often goes unrecognized. In fact, some perilunate dislocations (PLDs) or perilunate fracture-dislocations (PLFDs) may be missed in spite of critical clinical and radiographic examination, leading to a delay in treatment. If left untreated for an extended period of time the outcomes of surgical repair are significantly compromised. The recovery process is very long, often with poor prognosis (a high incidence of post-traumatic osteoarthritis and chronic wrist pain).

Early surgical management with the restoration of normal carpal anatomy is the gold standard for surgical repair of perilunate injuries. Surgical repair may involve an open reduction of the carpal bones, repair or reconstruction of the ligaments, and internal fixation of the fractures for PLDs and PLFDs. However, there is a huge variability with respect to approach and a lot to be desired with respect to outcomes. Open surgical procedures have been reported to lead to capsular scarring and joint stiffness and further interfere with the tenuous blood supply to the scaphoid and the torn ligaments. Another treatment options, which may aid in healing with reduced stiffness, is a combination of fluoroscopy and wrist arthroscopy which allows for anatomic reduction and fixation of the carpal bones with minimal tissue dissection. Injury variability and a wide array of surgical strategies make it difficult to treat and/or make improvements on specific techniques. Given the varied nature of the injury to this joint and varied outcomes, it is important to categorize the injury characteristics, the subsequent treatment options and the long-term outcomes of different clinical interventions. Many different surgical techniques have been advocated with a variety of reduction and fixation maneuvers, but unfortunately, the literature is sparse. There are disagreements with respect to volar, dorsal or combined surgical approaches. There is no consensus on the value of prophylactic carpal tunnel release. Some surgeons advocate direct ligament repair, while others feel it is unnecessary. A third group advocates for augmentation of the scapholunate ligament with screws or a graft. While most surgeons use smooth k-wires to hold the carpal reduction, there is no agreement on direction, number, size and position of k-wires. Further, there is no agreement on how long these k-wires should be left in place or on any aspect of rehabilitation.

Globally these injuries have been poorly studied and ideal timing for surgical intervention, optimal treatment and rehabilitation are unknown. The investigators hope to establish best-evidence clinical practice guidelines for the treatment of perilunate injuries including recommendations on the timing of reduction, the timing of surgery, best-practice surgical techniques and rehabilitation protocols. The C3PO Trial will represent the single largest prospective dataset ever accrued on perilunate injuries with the support of both Canadian hand and trauma-fellowshipped trained orthopaedic surgeons and corresponding research societies. This project has the potential to create a paradigm shift in the way surgeons think about the perilunate injuries from identification through to prognosis which would be beneficial to all orthopaedic traumatologists managing these patients.

The study has 3 major nested arms. The investigators have designed a national prospective registry intended to capture all perilunate injuries suffered in Canada over a 2 year period. Within this registry, the investigators have an embedded cohort to capture all injuries that present to registered trial centres. These patients will be consented to the cohort and subsequently have extensive perioperative data recorded as well as both short and long-term follow-up (with no modification of treatment). All data collection (i.e. relevant demographics, injury characteristics, surgical and management parameters) will be obtained and managed by a customized REDCap database housed at the trial coordinating centre. The third arm of this trial is a retrospective cohort in which patients previously treated for PLIs will be contacted as asked if they would be willing come back to clinic and be follow for the remaining period of the 10-year study.

Participants, 14 years of age or older, clinically diagnosed with a perilunate injury and willing to adhere to the study protocol will be included for study participation. They must be willing and able to attend all recommended post-operative follow-up visits based on the advice of their surgeon. All participants will complete questionnaires and undergo both clinical and radiographic evaluations. These evaluations will begin at baseline, continue at the first post-operative visit, and the following intervals: 3, 6, 12, 24, 60 and 120 months. Individuals will be excluded if they have cognitive impairment or unable to understand what participation in this study entails, a known alcohol or drug abuser, or anticipated to be non-compliant. The investigators anticipate overall 150 patients entered into the cohort, an additional 150 in the registry arm, and 150 patients identified retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 14 years of age or older
* The subject has been clinically diagnosed with a perilunate injury
* The subject is willing to adhere to the study protocol including required post-operative therapy, all scheduled follow-up visits, evaluations, and questionnaires (if applicable).

Exclusion Criteria:

There will be no limiting exclusion criteria.

Ages: 14 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who sustain a perilunate spectrum injury including dislocation and/or fracture.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) | Enrollment - 10 years
  The upper extremity scoring scale DASH is a validated tool for disorders of the elbow with a range from 0 (least disability) to 100 (most disability). Ten is the average score in the general population and the minimal clinically important difference (MCID) is 10. DASH contains 30 questions asking participants about their ability to perform activities and their symptoms. Each question ranges from 1 (no difficulty) to 5 (unable). There is also optional work and sports/performing arts modules.

SECONDARY OUTCOMES:
Radiographs | Enrollment - 10 years
  Radiographic evaluation for fracture healing and/or nonunion, and the number of participants requiring re-operation for contracture and also composite re-operation for all perilunate fractures and/or dislocations related causes. This will be completed by a radiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Neil J White, MD, FRCSC, Principal Investigator — University of Calgary
Locations (1):
- South Health Campus, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Garg B, Goyal T, Kotwal PP. Triple jeopardy: transscaphoid, transcapitate, transtriquetral, perilunate fracture dislocation. J Orthop Traumatol. 2013 Sep;14(3):223-6. doi: 10.1007/s10195-012-0195-x. Epub 2012 Apr 4. PMID 22476357
- [Background] Massoud AH, Naam NH. Functional outcome of open reduction of chronic perilunate injuries. J Hand Surg Am. 2012 Sep;37(9):1852-60. doi: 10.1016/j.jhsa.2012.06.009. Epub 2012 Jul 31. PMID 22854256
- [Background] Vitale MA, Seetharaman M, Ruchelsman DE. Perilunate dislocations. J Hand Surg Am. 2015 Feb;40(2):358-62; quiz 362. doi: 10.1016/j.jhsa.2014.10.006. Epub 2014 Nov 15. No abstract available. PMID 25459380
- [Background] Stanbury SJ, Elfar JC. Perilunate dislocation and perilunate fracture-dislocation. J Am Acad Orthop Surg. 2011 Sep;19(9):554-62. doi: 10.5435/00124635-201109000-00006. PMID 21885701
- [Background] Capo JT, Corti SJ, Shamian B, Nourbakhsh A, Tan V, Kaushal N, Debkowska M. Treatment of dorsal perilunate dislocations and fracture-dislocations using a standardized protocol. Hand (N Y). 2012 Dec;7(4):380-7. doi: 10.1007/s11552-012-9452-y. PMID 24294157
- [Background] Kozin SH. Perilunate injuries: diagnosis and treatment. J Am Acad Orthop Surg. 1998 Mar-Apr;6(2):114-20. doi: 10.5435/00124635-199803000-00006. PMID 9682074
- [Background] Perron AD, Brady WJ, Keats TE, Hersh RE. Orthopedic pitfalls in the ED: lunate and perilunate injuries. Am J Emerg Med. 2001 Mar;19(2):157-62. doi: 10.1053/ajem.2001.21306. PMID 11239263
- [Background] Weil WM, Slade JF 3rd, Trumble TE. Open and arthroscopic treatment of perilunate injuries. Clin Orthop Relat Res. 2006 Apr;445:120-32. doi: 10.1097/01.blo.0000205889.11824.03. PMID 16601413
- [Background] Sotereanos DG, Mitsionis GJ, Giannakopoulos PN, Tomaino MM, Herndon JH. Perilunate dislocation and fracture dislocation: a critical analysis of the volar-dorsal approach. J Hand Surg Am. 1997 Jan;22(1):49-56. doi: 10.1016/S0363-5023(05)80179-0. PMID 9018612
- [Background] Adkison JW, Chapman MW. Treatment of acute lunate and perilunate dislocations. Clin Orthop Relat Res. 1982 Apr;(164):199-207. PMID 7067286
- [Background] Souer JS, Rutgers M, Andermahr J, Jupiter JB, Ring D. Perilunate fracture-dislocations of the wrist: comparison of temporary screw versus K-wire fixation. J Hand Surg Am. 2007 Mar;32(3):318-25. doi: 10.1016/j.jhsa.2007.01.008. PMID 17336837
- [Background] Muppavarapu RC, Capo JT. Perilunate Dislocations and Fracture Dislocations. Hand Clin. 2015 Aug;31(3):399-408. doi: 10.1016/j.hcl.2015.04.002. PMID 26205701
- [Background] Hildebrand KA, Ross DC, Patterson SD, Roth JH, MacDermid JC, King GJ. Dorsal perilunate dislocations and fracture-dislocations: questionnaire, clinical, and radiographic evaluation. J Hand Surg Am. 2000 Nov;25(6):1069-79. doi: 10.1053/jhsu.2000.17868. PMID 11119665
- [Background] Krief E, Appy-Fedida B, Rotari V, David E, Mertl P, Maes-Clavier C. Results of Perilunate Dislocations and Perilunate Fracture Dislocations With a Minimum 15-Year Follow-Up. J Hand Surg Am. 2015 Nov;40(11):2191-7. doi: 10.1016/j.jhsa.2015.07.016. Epub 2015 Aug 29. PMID 26328900
- [Derived] Mitchell EC, Tottenham I, Grewal R, Curran MWT, White NJ. The Canadian Prospective Pragmatic Perilunate Outcomes (C3PO) trial; a protocol. BMC Musculoskelet Disord. 2025 Jan 31;26(1):93. doi: 10.1186/s12891-024-08227-x. PMID 39891160